CLINICAL TRIAL: NCT03910985
Title: Assessment of Reactance Parameters Measured by the Forced Oscillation Technique for the Bronchodilator Response in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire UCLouvain Namur (Other)
Responsible Party: Principal Investigator, Marchand Eric, Principal investigator Eric MARCHAND, Centre Hospitalier Universitaire UCLouvain Namur
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B039201938727
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Duovent HFA — bronchodilation

SUMMARY:
The aims of this study is :

* to assess the bronchodilator (DUOVENT HFA) response of parameters measured by the forced oscillations (FOT) and in particular the reactance parameters related to the presence of a limitation of expiratory flows
* to compare the response of the reactance parameters to bronchodilators with the conventional spirometric parameters (FEV1) and inspiratory capacity (IC), and according to the severity of the disease
* to assess and compare the relationship between the response to bronchodilators in terms of IC on the one hand and on the other hand in terms of FEV1, reactance parameters (measured by FOT), resistance parameters (measured by plethysmography and FOT)
* Assess and compare the relationship between dyspnea intensity assessed by various scales and conventional respiratory function parameters (spirometry, plethysmography, diffusion indices) and parameters measured by FOT

DETAILED DESCRIPTION:
Different techniques will be used during this study :

First, the FOT. The measurements will be performed using a Tremoflo-type (Thorasys Thoracic Medical System Inc.) device that generates an oscillating pressure waveform and measures impedance of the respiratory system and its components (resistance and reactance) as a function of frequency, as well as the respiratory system resonant frequency. Measurements will be performed during tidal breathing, the subjects breathing through the pneumotachograph of the system, with nose occluded, the cheeks supported by the hands (of the subjects or of an operator) to reduce the influence of the compliant upper airways. Three measurements of minimum 20 seconds duration will be recorded in the sitting position.

Second, the spirometry. The measurements will be carried out using a Medisoft Exp'air type of equipment. The parameters will be successively measured in the sitting position :

* The inspiratory capacity (IC) will be measured by maximal inspiratory maneuver starting from the functional residual capacity
* The thoracic gas volume (TGV), total lung capacity (TLC), as well as the airway resistance will be measured by plethysmography
* The diffusion indices (CO transfer factor (DL,CO) and CO transfer coefficient (KCO)) will be measured in apnea
* A spirometry will then be carried out. Three maneuvers with acceptability and reproducibility criteria will be performed

All these measurements will be carried out before the administration of the bronchodilator and 30 minutes after the administration of the bronchodilator (4 puffs of DUOVENT HFA, using an inhalation chamber).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD confirmed by post-bronchodilator (DUOVENT HFA 4 puffs) obstructive airway obstruction (FEV1/Forced Vital Capacity < Percentile 5) persisting after bronchodilatation
* Former or active smoking > 10 packs/year
* Age > 40 years
* Informed consent

Exclusion Criteria:

* Inability to comply with bronchodilator weaning time :

  6 hours for short-acting bronchodilators ; 12 hours for long-acting bronchodilators ; 24 hours for very long-acting bronchodilators
* Inability to comply with the 4 hours of smoking cessation before the measurements
* Inability to perform respiratory function tests
* Continuous oxygen therapy
* Close angle glaucoma
* History of urinary retention (only for patients not usually treated with anticholinergic bronchodilators)
* Pregnancy
* Acute illness contraindicating the performance of respiratory tests

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-04-23 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute inspiratory capacity increase | 30 minutes

IPD SHARING:
Plan to Share IPD: No